CLINICAL TRIAL: NCT00899002
Title: Molecular Analysis of Liver Cancer
Brief Title: Biomarkers in Stored Tumor Samples From Younger Patients With Liver Cancer
Status: Withdrawn | Type: Observational
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura W. Goff, MD, Assistant Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GI 0611; VU-VICC-GI-0611; VU-VICC-060479
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Liver Cancer
Keywords: childhood hepatocellular carcinoma; childhood liver cancer; adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Comparative Genomic Hybridization; Genetic Testing; Polymerase Chain Reaction; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from the tissue samples and analyzed for molecular signatures, i.e., genomic and proteomic analyses.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: comparative genomic hybridization
  Other Names: None specified
Genetic: molecular genetic technique
  Other Names: none noted
Genetic: mutation analysis
  Other Names: none noted
Genetic: polymerase chain reaction — Not noted
  Other Names: none specified
Genetic: proteomic profiling
  Other Names: none noted
Other: immunohistochemistry staining method — not noted
  Other Names: none specified
Other: laboratory biomarker analysis — not noted
  Other Names: none specified
Other: mass spectrometry — not noted
  Other Names: none specified
Other: medical chart review — not noted
  Other Names: none specified

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at biomarkers in stored tumor samples from younger patients with liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To characterize, at a molecular level, archived samples of tissue from young patients with fibrolamellar carcinoma and hepatocellular carcinoma in non-cirrhotic livers matched for age and sex.
* To perform genomic analysis on these tissue samples using array comparative genomic hybridization.
* To perform targeted gene mutation analysis on these samples by PCR.
* To perform proteomic profiling on fixed tissues in these samples by various proteomic methods, including IHC and mass spectrometry.
* To look for association between molecular aberrations and clinicopathologic features in these samples.

OUTLINE: Archived tissue samples are collected from the pathology department at Vanderbilt University Medical Center and from the Mayo Clinic in Rochester, Minnesota. Tissue samples are analyzed by genomic analysis using array comparative genomic hybridization, target gene mutation analysis by PCR, and proteomic profiling on fixed tissues using various proteomic methods, including IHC and mass spectrometry. Samples are also examined for association between molecular aberrations and clinicopathologic features found in each disease.

Clinical patient data (i.e., age, sex, race, date of diagnosis, risk factors, histology, surgical staging, follow-ups, date of death, and adjuvant therapy) are also collected.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of fibrolamellar carcinoma or hepatocellular carcinoma in a non-cirrhotic liver
* Archived tumor specimens available for analysis from Vanderbilt University or Mayo Clinic

Exclusion Criteria:

* Not specified

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample collection: 20 cases of fibrolamellar carcinoma and 20 hepatocellular carcinomas.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Identification of proteomic profiles and molecular pathways involved in tumor progression | After collection of tissue samples
  Genomic analysis, targeted gene mutation analysis, immunohistochemistry, and mass spectrometry will be employed to identify proteomic profiles and specific molecular pathways involved in tumor progression of fibrolamellar carcinoma and hepatocellular carcinoma

SECONDARY OUTCOMES:
Association between fibrolamellar carcinoma and hepatocellular carcinoma in terms of molecular aberrations and clinicopathologic features | After molecular analysis of tissue and after collection of clinicopathologic data
  Compare and contrast fibrolamellar carcinoma with hepatocellular carcinoma in terms of the molecular differences, tissue pathologies, and medical histories.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goff, MD, Study Chair — Vanderbilt-Ingram Cancer Center